CLINICAL TRIAL: NCT04138381
Title: A Multicenter, Phase Ib/II Trial of Selinexor as a Single Agent and in Combination With Imatinib in Patients With Metastatic and/or Unresectable Gastrointestinal Stromal Tumors (GISTs)
Brief Title: Selinexor as Single Agent and With Imatinib in Metastatic and/or Unresectable Gastrointestinal Stromal Tumors (SeliGIST)
Acronym: SeliGIST
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Grupo Espanol de Investigacion en Sarcomas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEIS 41; 2017-004761-28 (EudraCT Number)
Record Dates: First submitted 2019-09-16; First posted 2019-10-24 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Maximum Tolerated Dose; GIST; Metastatic Adult Soft Tissue Sarcoma; Drug Toxicity; Drug Use
Keywords: GIST; MTD; Imatinib; Selinexor; Phase Ib; Phase II; Unresectable; Metastatic
MeSH Terms: conditions — Sarcoma; Drug-Related Side Effects and Adverse Reactions; Neoplasm Metastasis | interventions — selinexor; Drug Combinations; Pharmaceutical Preparations; Imatinib Mesylate

STUDY DESIGN:
Intervention Model Description: Phase Ib/II, single-arm, two-cohort, non-randomized, open-label, multicenter, national clinical trial, single agent, combinations products
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- selinexor as a single agent and in combination with imatinib (Other): This is a single-arm, two-cohort, open label phase Ib/II trial studying the combination of oral imatinib 400 mg, once daily, and oral selinexor given once weekly (Cohort A); and single-agent oral selinexor 60 mg BIW (Cohort B). The study will consist of:
  * Cohort A: an initial escalation phase (Ib) evaluating increasing doses of selinexor in combination with fixed doses of imatinib administered in repeated 28-day cycles in advanced/metastatic, imatinib-resistant GIST patients, followed by en expansion phase (II) testing for safety and preliminary evidence of antitumor activity
  * Cohort B: single-agent, fixed selinexor dose in the same target population
  Interventions: Drug: Selinexor; Drug: Imatinib

INTERVENTIONS:
Drug: Selinexor — oral selinexor given once weekly (Cohort A), oral selinexor given BIW (Cohort B)
  Other Names: Drug Combination; Single agent
Drug: Imatinib — imatinib 400 mg, once daily (Cohort A)
  Other Names: Drug Combination

SUMMARY:
This is a single-arm, two cohort, open label phase I/II clinical trial studying the combination of oral imatinib 400 mg, once daily, and oral selinexor given once weekly (Cohort A); and single-agent oral selinexor 60 mg BIW (Cohort B). The study will consist of:

* Cohort A: an initial escalation phase (Ib) evaluating increasing doses of selinexor in combination with fixed doses of imatinib administered in repeated 28-day cycles in advanced/metastatic, imatinib-resistant GIST patients, followed by an expansion phase (II) testing for safety and preliminary evidence of antitumor activity
* Cohort B: single-agent, fixed selinexor dose in the same target population

DETAILED DESCRIPTION:
Clinical Study Objectives:

Primary clinical study objective

Cohort A:

1.- To determine the maximum tolerated dose (MTD) and recommended phase II doses (RP2D) of selinexor in combination with imatinib among unresectable and/or metastatic GIST patients with prior failure to at least imatinib for advanced/metastatic disease.

Cohort B:

1. To evaluate the clinical benefit rate (CBR: CR+PR+SD ≥ 16 wks)

Secondary clinical study objectives (both cohorts A and B)

1. To evaluate the clinical benefit rate (CBR: CR+PR+ SD ≥ 16 wks)
2. To evaluate progression free survival (PFS)
3. To evaluate overall survival (OS)
4. To evaluate the objective response rate (ORR)
5. To evaluate the safety profile according to CTCAE 4.03
6. To compare PFS on selinexor and imatinib and on selinexor in monotherapy with PFS on last prior anti-cancer therapy.

Translational Study Objective - To explore the relationship between GIST genotype and CBR with selinexor and imatinib, and selinexor as single-agent

Pharmacokinetics Study Objective

- To measure the plasma concentration of imatinib and selinexor at limited timepoints specificed in schedule of assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of study entry.
2. Histologically confirmed metastatic and/or unresectable GIST. Patients must demonstrate prior failure to at least imatinib. Any number of previous therapies for GIST is allowed.
3. Failure of imatinib is defined as disease progression after ≥ 6 months of treatment with imatinib for advanced/metastatic disease. Exception to this rule is GIST patients with documented KIT or PDGFRA mutations.
4. Measurable disease per modified RECIST 1.1.
5. ECOG performance status 0 to 2.
6. Adequate hematopoietic function (within 7 days prior to enrollment):

   1. Hemoglobin ≥ 9.0 g/dL (90 g/L).
   2. Absolute neutrophil count ≥ 1000/mm3.
   3. Platelets ≥ 100,000 /mm3. Patients must have at least a 2-week interval from the last red blood cell (RBC) transfusion and/or growth factor support prior to the Screening hemoglobin and neutrophil assessment. However, patients may receive RBC, growth factor support, and/or platelet transfusions as clinically indicated per institutional guidelines during the study.
7. Adequate organ function (within 7 days prior to enrollment):

   1. Alanine aminotransferanse (ALT) and aspartate aminotransferanse (AST)

      ≤2.5 x upper limit of normal (ULN), or ≤ 5.0 x ULN if liver metastases are present.
   2. Alkaline phosphatase (ALP) limit < 2.5 x ULN or ≤ 5.0 x ULN if liver metastases are present.
   3. Total serum bilirubin ≤ 2 x ULN. Patients with Gilbert's syndrome must have a total bilirubin of < 3 × ULN.
   4. Adequate renal function: estimated creatinine clearance of ≥ 30 mL/min, calculated using the formula of Cockroft and Gault
8. Patients must be able to swallow oral medication and no malabsorption condition.
9. Willingness to use effective means of birth control throughout the duration of clinical study and for at least 3 months after completion of study drug.
10. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of study drug administration.
11. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Cohort A: Intolerance to first-line treatment imatinib 400mg daily.
2. Use of any approved tyrosine kinase inhibitors or investigational agents within 1 week or 5 half-lives of the agent, whichever is shorter, prior to receiving study drugs.
3. Participants who have had radiotherapy within 4 weeks prior to study entry.
4. Major surgery or significant traumatic injury within 4 weeks prior to study entry.
5. Presence of symptomatic or uncontrolled brain or central nervous system metastases.
6. Known or suspected allergy or hypersensitivity to the selinexor, imatinib or any of its components.
7. Patient has a history of another primary malignancy that has been diagnosed or required therapy within 1 year prior to the first dose of study drug (The following are exempt from the 1-year limit: completely resected basal cell and squamous cell skin cancer, curatively treated localized prostate cancer, and completely resected carcinoma in situ of any site.)
8. Unstable cardiovascular function: • Symptomatic ischemia, or • Uncontrolled clinically significant conduction abnormalities (i.e., ventricular tachycardia on antiarrhythmic agents are excluded; 1st degree atrioventricular (AV) block or asymptomatic left anterior fascicular block/right bundle branch block (LAFB/RBBB) will not be excluded), or • Congestive heart failure (CHF) NYHA Class ≥ 3, or • Myocardial infarction (MI) within 3 months. • Left ventricular ejection fraction < 40 %. • Hypertension > 140 mm Hg systolic or > 90 mm Hg diastolic with or without antihypertensive therapy.
9. Ongoing infection > Grade 2.
10. Patients with any seizure disorder requiring medication.
11. HIV-positive individuals on combination antiretroviral.
12. Patients with active hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy.
13. Serious psychiatric or medical conditions that could interfere with treatment.
14. Pregnant or lactating females.
15. Strong CYP3A4 inhibitors (e.g. clarithromycin, indinavir, itraconazole, ketoconazole , nefazodone , nelfinavir , posaconazole, ritonavir, saquinavir, telithromycin, voriconazole) or strong CYP3A4 inducers (e.g. carbamazepine, phenobarbital, phenytoin, rifampin, St. John's Wort) within 28 days or 5 drug half-lives (if drug half-life in patients is known), whichever is longer, before start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-16 (Actual); Primary Completion 2023-04-16 (Estimated); Study Completion 2023-04-16 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) for the use of Imatinib in combination with Selinexor | 32 months
  Maximum tolerated dose (MTD) is defined as the highest dose level with ≤1 out of 6 patients experiencing a dose limiting toxicity (DLT) during the first 28 days of treatment. Dose escalation cohort (Phase 1b) seeks to determine the frequency and characteristics of DLTs of the selinexor plus imatinib combination at each dose level during the first cycle of therapy. Phase Ib will be carried out in standard 3+3 format, based on the toxicities found during the first cycle of therapy.
Clinical benefit rate (CBR) for the use of selinexor in monotherapy | 24 months
  Clinical benefit rate (CBR) is defined as CR+PR+SD ≥ 16 wks

SECONDARY OUTCOMES:
Progression free survival (PFS) | 32 months
  Efficacy measured by PFS assessed by median time. PFS is defined as the time between the date of first experimental treatment dose and the date of disease progression (according to RECIST 1.1 criteria).
Overall survival (OS) | 32 months
  Efficacy measured by OS. OS is defined as the time between the date of first experimental treatment dose and the date of death due to any cause. OS will be censored on the last date a subject was known to be alive, or when the last enrolled patiens are followed up to for 12 months, whichever is early.
Objective response rate (ORR) | 32 months
  Efficacy measured by ORR. ORR is defined as the number of subjects with a best overall response (BOR) of complete response (CR) or partial response (PR) divided by the number of response evaluable subjects (according to RECIST 1.1 and Choi criteria).
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 32 months
  Safety profile of the experimental treatment, through assessment of adverse event type, incidence, severity, time of appearance, related causes, as well as physical explorations and laboratory tests. Number of participants with treatment-related adverse events as assessed by CTCAE v4.03.
  Toxicity will be graded and tabulated by using CTCAE 4.03.
GIST genotype and CBR with selinexor and imatinib (Translational) Study Objective | 32 months
  GIST genotype determinations and its correlation with response to the treatment with selinexor and imatinib in terms of clinical benefit (CBR).
Measure the plasma concentration of imatinib and selinexor (Pharmacokinetics)Study Objective | 32 months
  To measure the plasma concentration of imatinib and selinexor at limited timepoints specificed in schedule of assessment.
Clinical benefit rate (CBR) | 24 months
  Number of patient with CBR ≥ 30% lasting ≥ 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Serrano, MD, Principal Investigator — Hospital Vall d´Hebron
Locations (6):
- Spain (6):
  - Hospital Virgen del Rocio, Seville, Andalusia
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - H Vall d'Hebrón, Barcelona, Catalonia
  - Hospital Miguel Servet, Zaragoza, Zaragoza, Aragón
  - Hospital La Paz, Madrid
  - Hospital Virgen de la Arrixaca, Murcia

IPD SHARING:
Plan to Share IPD: No
The final publication of the trial results will be written by the international coordinating investigators on the basis of the final analysis performed. The draft manuscript will be reviewed by the coordinating investigators and other co-authors. After revision the manuscript will be sent to a major scientific journal. Results obtained in the different strata may be separately published.